CLINICAL TRIAL: NCT06707909
Title: The Local Effect of Vitamin K2 on Bone Remodeling in Socket Preservation of Mandibular Single Rooted Teeth Randomized Clinical Trail
Brief Title: The Local Effect of Vitamin K2 on Bone Remodeling in Socket Preservation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hussien Mohamed Elsawaf, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Socket Preservation
MeSH Terms: interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menaquinone group (Active Comparator): Tooth extraction will perform under local anesthesia All sockets were thoroughly curetted to remove granulation tissue, followed by irrigation and rinsing with sterile saline. the socket will be filled with crushed capsule of vitamin k2(menaquinone) and cover with an absorbent sponge a Figure of eight tension-free non-resorbable 3-0 sutures will be placed over the filled socket to stabilize the graft material in the socket and to achieve soft tissue stability.
  Bone density and socket dimensions will be evaluated immediately after extraction with graft material and after 4 months by using a cone beam computed tomography (CBCT) radiograph and at the time of implant placement core biopsy will be taken for histomorphometric analysis.
  Interventions: Drug: Menaquinone
- control group (No Intervention): Tooth extraction will perform under local anesthesia All sockets were thoroughly curetted to remove granulation tissue, followed by irrigation and rinsing with sterile saline. the socket will be left to heal without grafting, and it will be covered with an absorbent sponge. A figure-of-eight tension-free non-resorbable 3-0 sutures will be placed over the socket.
  Bone density and socket dimensions will be evaluated immediately after extraction with graft material and after 4 months by using a cone beam computed tomography (CBCT) radiograph and at the time of implant placement core biopsy will be taken for histomorphometric analysis.

INTERVENTIONS:
Drug: Menaquinone — the socket will be filled with crushed capsule of vitamin k2 menaquinone in study group
  Other Names: vitamin k2 (Menaquinone)
  Arms: Menaquinone group

SUMMARY:
This study is a randomized controlled trial comparing the effects of socket grafting with crushed vitamin K2 (menaquinone)capsules versus no grafting on bone density and socket dimensions following tooth extraction. Patients are randomly assigned to one of two groups:

Study Group (Group I): Patients receive socket grafting with crushed vitamin K2 (menaquinone) capsules. The socket is covered with an absorbent sponge, and non-resorbable sutures are placed to stabilize the graft material and achieve soft tissue stability.

Control Group (Group II): Patients undergo socket healing without grafting. The socket is covered with an absorbent sponge, and non-resorbable sutures are placed over it.

Outcome measures include bone socket dimensions evaluated immediately after extraction with graft material, as well as assessment after 4 months using cone beam computed tomography (CBCT) radiographs. Additionally, core biopsies are taken at the time of implant placement.

DETAILED DESCRIPTION:
The study is designed as a randomized controlled trial to investigate the effects of socket grafting with crushed vitamin K2 (menaquinone) capsules compared to no grafting on bone density and socket dimensions following tooth extraction.

Participants: Patients scheduled for tooth extraction are enrolled in the study and randomized into two equal groups.

11. Interventions

- Patients were randomly divided into two equal groups.

In both groups:

Tooth extraction will perform under local anesthesia All sockets were thoroughly curetted to remove granulation tissue, followed by irrigation and rinsing with sterile saline.

Bone density and socket dimensions will be evaluated immediately after extraction with graft material and after 4 months by using a cone beam computed tomography (CBCT) radiograph and at the time of implant placement core biopsy will be taken.

In group I (study): the socket will be filled with crushed capsule of vitamin k211. Interventions

- Patients were randomly divided into two equal groups.

In both groups:

Tooth extraction will perform under local anesthesia All sockets were thoroughly curetted to remove granulation tissue, followed by irrigation and rinsing with sterile saline.

Bone density and socket dimensions will be evaluated immediately after extraction with graft material and after 4 months by using a cone beam computed tomography (CBCT) radiograph and at the time of implant placement core biopsy will be taken.

In group I (study): the socket will be filled with crushed capsule of vitamin k2 and cover with an absorbent sponge a Figure of eight tension-free non-resorbable 3-0 sutures will be placed over the filled socket to stabilize the graft material in the socket and to achieve soft tissue stability.

in group II (control): the socket will be left to heal without grafting, and it will be covered with an absorbent sponge. A figure-of-eight tension-free non-resorbable 3-0 sutures will be placed over the socket.

and cover with an absorbent sponge a Figure of eight tension-free non-resorbable 3-0 sutures will be placed over the filled socket to stabilize the graft material in the socket and to achieve soft tissue stability.

in group II (control): the socket will be left to heal without grafting, and it will be covered with an absorbent sponge. A figure-of-eight tension-free non-resorbable 3-0 sutures will be placed over the socket.

ELIGIBILITY:
Inclusion Criteria:• Age > 18 years without other age or gender restrictions.

* Patients requiring extraction of mandibular single-rooted teeth.

Exclusion Criteria:

* • Patients with systemic conditions affecting bone metabolism.

  * Allergies or sensitivities to hydroxyapatite or Vitamin K2
  * Untreated or residual periodontal disease;
  * Uncontrolled diabetes (HbA1c > 7.5%);
  * Head and/or neck radiotherapy
  * Immunosuppressive therapy
  * Pregnant or nursing
  * Substance abuse
  * Treated or under treatment with intravenous amino-bisphosphonates
  * Patients participating in other studies, if the present protocol could not be properly followed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss | baseline and 4 month after extraction
  At the time of extraction, CBCT imaging will provide baseline data on the initial bone structure This baseline measurement serves as a reference point for evaluating any subsequent changes in bone density and morphology.
  After four months, another CBCT scan will be conducted to assess the amount of marginal bone loss that has occurred since the initial extraction. By comparing the post-extraction CBCT images with those taken after four months, researchers can quantify any changes in bone volume and identify any areas of concern related to bone resorption. The unit of measurement for the primary outcome, vertical bone change (socket height), is millimeters (mm).

SECONDARY OUTCOMES:
Primary stability | at time of implant placment
  For the primary stability assessment, the Implant Stability Quotient (ISQ) will be utilized. ISQ is a non-invasive and widely used method for evaluating the initial stability of dental implants during placement. Unit of Measurement: Implant Stability Quotient (ISQ)
amount of new bone formation | baseline and 4 month after extraction
  amount of new bone formation," histomorphometric analysis will be employed. This method involves the microscopic examination and quantification of bone tissue characteristics to assess the extent of bone formation.
  Histomorphometric analysis allows researchers to evaluate the quality and quantity of newly formed bone in the extraction site or implantation site. It involves taking tissue samples (biopsies) from the area of interest and then processing these samples for microscopic examination. Unit of Measurement: Bone area percentage (%)

OTHER OUTCOMES:
Secondary stability | 4 month post-implant placement
  the Implant Stability Quotient (ISQ) will be utilized. ISQ is a non-invasive and widely used method for evaluating the stability. Unit of Measurement: Implant Stability Quotient (ISQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo, Cairo, Cairo Governorate, Egypt